CLINICAL TRIAL: NCT06880341
Title: MagNETs- Managing Transient Neurologic Episodes in Surgery for Moyamoya Disease
Brief Title: Managing Transient Neurologic Episodes in Surgery for Moyamoya Disease
Acronym: MagNETs
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Gary Steinberg, MD, PhD, Professor and Former Chair, Department of Neurosurgery, School of Medicine, Stanford University
Other Study IDs: 77828
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Moya Moya Disease
MeSH Terms: conditions — Moyamoya Disease | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- MoyaMoya Subjects: Subjects will receive standard of care moyamoya surgical intervention and be followed for 30 days post for transient neurological episodes (TNEs).
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — Standard of care treatment of Transient Neurologic Events (TNEs) as needed

SUMMARY:
The goal of this study is to study the incidence of post-operative Transient Neurologic Events (TNEs) within 30 days postoperatively, as assessed by clinical neurological scales, binned by week. Collect data on all interventions and assessments performed during the recovery post surgery up to 30 days, to understand what factors might cause Transient Neurologic Events (TNEs) and determine how these can be reduced in Moyamoya subjects post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Moyamoya Disease (MMD) patients undergoing direct extracranial-intracranial (ECIC) bypass. Patients above the age of 3 years old are eligible for the study

Exclusion Criteria:

* Renal dysfunction, electrolyte disturbances neuromuscular disorders including Myaesthenia Gravis, heart block

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Moyamoya subject undergoing a standard of care direct and indirect extracranial-intracranial (ECIC) bypass.
Sampling Method: Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Transient Neurologic Events (TNEs) | 30 days post-surgery
  Number of Incidence of post-operative Transient Neurologic Events (TNEs) within 30 days postoperatively, as assessed by clinical neurological scales (e.g., NIH Stroke Scale, Modified Rankin Scale), binned by week.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No